CLINICAL TRIAL: NCT05491655
Title: High Intensity His Bundle Pacing in Heart Failure Patients With Narrow QRS Outcome Study
Acronym: HIPPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Grigorios Katsouras, Cardiologist, Principal Investigator, Miulli General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGH_003
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Conduction System; His Bundle Pacing; Heart Failure; Cardiomyopathies
Keywords: His bundle pacing; conduction system pacing; Heart failure; Cardiomyopathy; narrow QRS; Ejection Fraction
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects will be blinded to treatment arm. Echocardiographic evaluation will be performed by study physician blinded to lead placement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity His bundle pacing (Experimental): After implantation of the device there will be a 1-month run-in period that the device will be programmed to deliver His bundle pacing therapy during this period at 3.5V/1msec.
  After one month these patients will continue to receive active pacing treatment with 3.5V/1msec.
  Interventions: Device: High Intensity His Bundle pacing
- Back up only ventricular pacing (Sham Comparator): After implantation of the device there will be a 1-month run-in period that the device will be programmed to deliver His bundle pacing therapy during this period at 2V/1msec.
  After one month these patients will receive back up only pacing (pacemaker programmed to VVI 30 bpm or AAI(R)-DDD(R) 50bpm) for 6 months.
  Interventions: Device: High Intensity His Bundle pacing

INTERVENTIONS:
Device: High Intensity His Bundle pacing — All patients will be implanted with an Implantable cardioverter defibrillator (ICD) and an ICD lead in the right ventricle (either RV apex or RV septum). In all patients a pacing lead will be positioned in the right atrium (typically the right atrial appendage). All patients will have a pacemaker lead positioned on the His bundle to obtain direct His-bundle capture.

SUMMARY:
Cardiac Resynchronization Therapy (CRT) decreases heart failure hospitalizations and mortality and increases left ventricular Ejection Fraction (EF) in patients with dilated cardiomyopathy, left bundle branch block and QRS duration >130msec. His bundle pacing has a similar effect in this category of patients. However, CRT is not beneficial in heart failure (HF) patients with narrow QRS. His-bundle pacing delivers physiological ventricular activation and has been shown to improve acute hemodynamic function in patients with heart failure, a prolonged PR interval, and either a narrow QRS or RBBB through AV delay optimization. We observed an acute hemodynamic effect during application of higher pacing output (3.5 Volts/1 msec) in HF patients with dilated or ischemic cardiomyopathy and narrow QRS independently of the paced QRS duration or AV delay shortening.

This is a single-center, prospective randomized single-blinded study, recruiting a sub-population of patients with heart failure (dilated or ischemic cardiomyopathy, EF<50%, narrow QRS (<110 msec), in optimal medical treatment who have an indication for ICD.

DETAILED DESCRIPTION:
Cardiac Resynchronization Therapy (CRT) decreases heart failure hospitalizations and mortality and increases left ventricular Ejection Fraction (EF) in patients with dilated cardiomyopathy, left bundle branch block and QRS duration >130msec. His bundle pacing has a similar effect in this category of patients. However, CRT is not beneficial in heart failure (HF) patients with narrow QRS. His-bundle pacing delivers physiological ventricular activation and has been shown to improve acute hemodynamic function in patients with heart failure, a prolonged PR interval, and either a narrow QRS or Right Bundle Branch Block (RBBB) through atrioventricular (AV) delay optimization. We observed an acute hemodynamic effect during application of higher pacing output (3.5 Volts/1 msec) in HF patients with dilated or ischemic cardiomyopathy and narrow QRS independently of the paced QRS duration or AV delay shortening.

This is a single-center, prospective randomized single-blinded study, recruiting a sub-population of patients with heart failure (dilated or ischemic cardiomyopathy, EF<50%, narrow QRS (<110 msec), in optimal medical treatment who have an indication for ICD.

All patients will be implanted with a CRT (Cardiac Resynchronization Therapy) defibrillator with one of the leads positioned on the His bundle to obtain direct His-bundle capture. (There will be a 1-month run-in period where the output voltage will be 3.5 Volts/1 or 2V/1msec according to the group so as to obtain stable threshold).

A single-blinded design will then be employed to investigate the effect of His bundle pacing. Patients will be allocated in random order to six-month treatment periods in each of the following two states (1) 3.5 Volts/1 msec pacing output direct His-bundle pacing, AV delay will be programmed in order to obtain a PR interval of 120-140msec; (2)back up only pacing (pacemaker programmed to VVI 30 bpm or AAI(R-DDD(R) 60bpm). Endpoint measurements will be taken at baseline, 1 month run-in period of 3.5 Volts/1 msec or 2V/1msec pacing output and 6 months post randomization. Treating Physicians will be aware of assignment in order to facilitate routine device follow-up. Echocardiographic and electrocardiographic evaluation will be performed in a blinded manner. Treatment allocation will be blinded to the endpoint assessor and the patient.

Patients entering the study will attend for implantation of a CRT pacemaker device with one lead positioned on the His bundle. This will be performed in Miulli General Hospital (and other participating centres) no later than 2 months after the patient's screening visit.

Before the intervention patients will be randomized to either receive active pacing treatment with 3.5 V/1 msec or back up only pacing (pacemaker programmed to VVI 30 bpm or AAI(R)-DDD(R) 60) for 6 months. All patients will be implanted with an Implantable cardioverter defibrillator (ICD) and an ICD lead in the right ventricle (RV) (either RV apex or RV septum). In all patients a pacing lead will be positioned in the right atrium (typically the right atrial appendage). All patients will have a pacemaker lead positioned on the His bundle to obtain direct His-bundle capture.

After implantation of the device there will be a 1-month run-in period that the device will be programmed to deliver His bundle pacing therapy during this period at 3.5 Volts/1msec or 2V/1msec according to the assignment group.

One month after patients are implanted with their device, patients will either receive active pacing treatment with 3.5 V/1 msec or back up only pacing (pacemaker programmed to VVI 30 bpm or AAI(R)-DDD(R) 60bpm) for 6 months. Treatment allocation will be obtained using an Interactive Web Response System (IWRS) programmed with a randomization schedule provided by the trial statistician. Appropriate blocking will be used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Ventricular Ejection Fraction (EF) < 50%; BNP needs to be ≥250ng/L or N Terminal-pro BNP≥600ng/L for patients with EF 36-50% and they should have an ICD indication
* New York Heart Association (NYHA) class I-IV
* Narrow QRS duration (≤110ms) on 12 lead ECG

Exclusion Criteria:

* Other serious medical condition with life expectancy of less than 1 year
* Lack of capacity to consent
* Pregnancy
* Previous aortic valve surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | Baseline pre-intervention, randomisation and 6 months post randomisation
  change in left ventricular ejection fraction measured by 2D echo at 6 months compared to baseline

SECONDARY OUTCOMES:
Changes in B-type Natriuretic Peptide (BNP) | Baseline pre-intervention, randomisation and 6 months post randomisation
  Measured from blood samples
Changes in Quality of Life (QOL) Scores | Baseline pre-intervention,1 and 6 months post randomisation
  Change in QOL measured by the Kansas City Cardiomyopathy Questionnaire at 1 and 6 months compared to baseline. Scores are scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest
Changes in arrhythmia burden | 1 month and 6 months post randomization.
  Measured during Pacemaker control

CONTACTS AND LOCATIONS:
Locations (1):
- Miulli General Hospital, Acquaviva delle Fonti, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigorios E Katsouras, Stavros Stavrakis, Beneficial effects of high output His bundle pacing in patients with heart failure and narrow QRS, Heart Rhythm, Vol 20, Issue 5, Supplement, S479-S480
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Upadhyay GA, Vijayaraman P, Nayak HM, Verma N, Dandamudi G, Sharma PS, Saleem M, Mandrola J, Genovese D, Tung R; His-SYNC Investigators. His Corrective Pacing or Biventricular Pacing for Cardiac Resynchronization in Heart Failure. J Am Coll Cardiol. 2019 Jul 9;74(1):157-159. doi: 10.1016/j.jacc.2019.04.026. Epub 2019 May 9. No abstract available. PMID 31078637
- [Background] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Background] Whinnett ZI, Shun-Shin MJ, Tanner M, Foley P, Chandrasekaran B, Moore P, Adhya S, Qureshi N, Muthumala A, Lane R, Rinaldi A, Agarwal S, Leyva F, Behar J, Bassi S, Ng A, Scott P, Prasad R, Swinburn J, Tomson J, Sethi A, Shah J, Lim PB, Kyriacou A, Thomas D, Chuen J, Kamdar R, Kanagaratnam P, Mariveles M, Burden L, March K, Howard JP, Arnold A, Vijayaraman P, Stegemann B, Johnson N, Falaschetti E, Francis DP, Cleland JGF, Keene D. Effects of haemodynamically atrio-ventricular optimized His bundle pacing on heart failure symptoms and exercise capacity: the His Optimized Pacing Evaluated for Heart Failure (HOPE-HF) randomized, double-blind, cross-over trial. Eur J Heart Fail. 2023 Feb;25(2):274-283. doi: 10.1002/ejhf.2736. PMID 36404397